CLINICAL TRIAL: NCT00097981
Title: A Randomized, Open-Label, Multi-Center Trial Comparing Thalidomide Plus Dexamethasone (Thal-Dex) Versus DOXIL plusThalidomide Plus Dexamethasone (DOXIL -Thal-Dex) in Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Thalidomide Plus Dexamethasone (Thal-Dex) Versus DOXIL plusThalidomide Plus Dexamethasone (DOXIL -Thal-Dex) in Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004579; DO04-23-006 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Results first posted 2008-11-27 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Newly diagnosed multiple myeloma; Thalidomide; Dexamethasone; DOXIL; Pegylated liposomal hydrochloride doxorubicin injection
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide + dexamethasone (Active Comparator)
  Interventions: Drug: Thalidomide; Drug: Dexamethasone
- Thalidomide + dexamethasone + DOXIL (Experimental)
  Interventions: Drug: Thalidomide; Drug: Dexamethasone; Drug: DOXIL

INTERVENTIONS:
Drug: Thalidomide — Participants will receive thalidomide orally every night (at bedtime) without food on days 1-28 and dosing will gradually increase during Cycle 1 starting at 50 mg on 1 to 7 days, 100 mg on 8 to 14 days, 150 mg on 15 to 21 days, and 200 mg 22 to 28 days. Thalidomide 200 mg per day will be administered for subsequent cycles. Participants will receive thalidomide for minimum of 4 cycles and a maximum of 12 cycles.
Drug: Dexamethasone — Participants will receive dexamethasone 40 mg orally on Days 1 to 4, 9 to 12 and 17 to 20.
Drug: DOXIL — DOXIL 40 mg/m2 will be administered iintravenously (into a vein) on Day 1.
  Arms: Thalidomide + dexamethasone + DOXIL

SUMMARY:
The purpose of this study is to determine if Thalidomide + Dexamethasone or DOXIL (doxorubicin HCl liposome injection) + Thalidomide + Dexamethasone is more effective in treating newly diagnosed patients with multiple myeloma. The number of patients whose multiple myeloma disappears for a period of time (complete Response) will be studied to make the determination of which treatment is more effective.

DETAILED DESCRIPTION:
This is a multi-center, open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance) study to compare the safety and effectiveness of Thalidomide + Dexamethasone versus DOXIL (doxorubicin HCl liposome injection) + Thalidomide + Dexamethasone in patients with newly diagnosed multiple myeloma. Treatments are administered in 28-day cycles. Patients will receive 4 to 12 treatment cycles, depending on the response of their multiple myeloma to the treatment (measured according to the European Group for Blood and Marrow Transplant Response Criteria). Patients will have additional tests that include Multiple Gated Acquisition (MUGA) scans or echocardiograms to assess the patients for potential cardiotoxicity that could be related to treatment with DOXIL (doxorubicin HCl liposome injection). Maximum duration of study participation for each participant will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed multiple myeloma (per International Myeloma Working Group [IMWG] criteria
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Adequate absolute neutrophil count (ANC), platelet count and hemoglobin
* Adequate serum calcium
* Enrollment in System for Thalidomide Education and Prescribing Safety Program (S.T.E.P.S.)

Exclusion Criteria:

* No treatment with dexamethasone for multiple myeloma
* No peripheral neuropathy of Grade 2 or higher
* No Left Ventricular Ejection Fraction (LVEF) of less than 45 percentage
* No history of life-threatening thromboembolic events of any kind (ie, myocardial infarction, pulmonary embolism, stroke or others), within 1 year before enrollment in the study
* No deep vein thrombosis (DVT) within 1 year of enrollment
* No current anticoagulation for DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (58):
- United States (58):
  - Fountain Valley, California
  - Greenbrae, California
  - La Verne, California
  - Los Angeles, California
  - Denver, Colorado
  - New London, Connecticut
  - Boca Raton, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orange City, Florida
  - Ormond Beach, Florida
  - Lawrenceville, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Minneapolis, Minnesota
  - Saint Louis Park, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Jersey City, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - Armonk, New York
  - Box 302, New York
  - Brooklyn, New York
  - Nyack, New York
  - The Bronx, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Pittsburgh, Pennsylvania
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Easley, South Carolina
  - Sumter, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Bedford, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Fredericksburg, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Vancouver, Washington
  - Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 225 participants were randomnly assigned to treatment, 113 participants to the thal/dex group and 112 participants to the DOXIL/thal/dex group.
Groups:
- Thalidomide + Dexamethasone: Participants received thalidomide every night (at bedtime) without food on Days 1 to 28 and dosing was gradually increased during Cycle 1 starting at 50 mg on Days 1 to 7, 100 mg on Days 8 to 14, 150 mg on 15 to 21, and 200 mg on Days 22 to 28. Thalidomide 200 mg per day was administered for subsequent cycles. Dexamethasone 40 mg was administered by mouth on Days 1 to 4, 9 to 12 and 17 to 20.
- DOXIL + Thalidomide + Dexamethasone: DOXIL 40 mg/m2 was administered intravenously on Day 1 and thalidomide every night (at bedtime) without food on Days 1-28 and dosing was gradually increased during Cycle 1 starting at 50 mg on Days 1 to 7, 100 mg on Days 8 to 14, 150 mg on 15 to 21, and 200 mg on Days 22 to 28. Thalidomide 200 mg per day was administered for subsequent cycles. Dexamethasone 40 mg was administered by mouth on Days 1 to 4, 9 to 12 and 17 to 20.
Period: Overall Study
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Started | 113 (Enrollment at randomization) | 112 (Enrollment at randomization)
Received Study Medication | 110 | 106
Completed | 7 (Completion of 2 or more cycles after CR or nCR, or completion of 12 cycles.) | 12 (Completion of 2 or more cycles after CR or nCR, or completion of 12 cycles.)
Not Completed | 106 | 100
Not completed — Adverse Event | 31 | 44
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 2 | 4
Not completed — Physician Decision | 7 | 1
Not completed — Disease Progression | 8 | 2
Not completed — Transplant planned | 28 | 27
Not completed — Other | 19 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone | Total
Number analyzed (Participants) | 113 | 112 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.29 (10.31) | 60.62 (10.79) | 60.45 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 44 | 95
  Male | 62 | 68 | 130

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate: Number of Participants Who Achieved a Complete Response
Description: Complete response rate to study medication is defined as number of participants who acheived complete response by the local investigator according to the current European Group for Blood and Marrow Transplantation (EBMT) criteria. According to EBMT criteria, CR is defined as the absence of serum and urine monoclonal paraprotein + plus no increase in size or number of lytic bone lesions. Complete response was assessed at the beginning of every treatment cycle prior to treatment, starting at Cycle 2.
Time Frame: From Cycle 2 until 28 days following completion of treatment
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Number; unit: Participants
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Participants | 5 | 8
Statistical Analysis 1: Comparison: Thalidomide + Dexamethasone vs DOXIL + Thalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.49, Cochran-Mantel-Haenszel; Stratified by International Prognostic Index (IPI) stage 1,2 and 3

2. Secondary Outcome: Overall Response: Number of Participants Who Achieved a Complete Response (CR) or Partial Response (PR)
Description: Overall response to study medication is defined as number of participants who acheived a complete response (CR) or partial response (PR) by the local investigator according to the current European Group for Blood and Marrow Transplantation (EBMT) criteria. According to EBMT criteria, CR is defined as the absence of serum and urine monoclonal paraprotein + plus no increase in size or number of lytic bone lesions; and PR is defined as not all CR criteria + 50 percentage or more reduction in serum monoclonal paraprotein.
Time Frame: From Cycle 2 until 28 days following completion of treatment
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Number; unit: Participants
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Participants | 81 | 76
Statistical Analysis 1: Comparison: Thalidomide + Dexamethasone vs DOXIL + Thalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.42, Cochran-Mantel-Haenszel; Stratified by International Prognostic Index (IPI) stage 1,2 and 3

3. Secondary Outcome: Time to 1st Response
Description: Time to first response was defined as the interval from date of randomization to date of achieving a partial response (PR) or better according to the current European Group for Blood and Marrow Transplantation (EBMT) criteria. According to EBMT criteria, PR is defined as not all CR criteria + 50 percentage or more reduction in serum monoclonal paraprotein.
Time Frame: From Cycle 2 until 28 days following completion of treatment
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Days | 44 [37 to 58] | 58 [44 to 60]
Statistical Analysis 1: Comparison: Thalidomide + Dexamethasone vs DOXIL + Thalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.42, Log Rank

4. Secondary Outcome: Time to Progression
Description: Time to progression is the interval between the date of randomization until disease progression or death due to progression.
Time Frame: From randomization until death or as assessed up to 2 years post last participant last treatment visit
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Days | 584 [347 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of events observed by end of study. | 408 [350 to 597]
Statistical Analysis 1: Comparison: Thalidomide + Dexamethasone vs DOXIL + Thalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.5162, Log Rank

5. Secondary Outcome: Overall Survival: Number of Participants Died Due to Any Cause
Time Frame: From randomization until death or as assessed up to 2 years post last participant last treatment visit
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Number; unit: Participants
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Participants | 21 | 22
Statistical Analysis 1: Comparison: Thalidomide + Dexamethasone vs DOXIL + Thalidomide + Dexamethasone; Test type: Superiority or Other; p = 0.93, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 0.975, 95% CI 2-sided [0.529 to 1.797]

6. Secondary Outcome: Transplantation: Number of Participants Who Underwent Transplantation (Peripheral Stem Cell / Bone Marrow)
Time Frame: From randomization until death or as assessed up to 2 years post last participant last treatment visit
Population: Intent-to-treat: Participants who were randomized to receive the treatment.
Measure: Number; unit: Participants
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 112
Participants | 30 | 28

7. Secondary Outcome: Engraftment: Number of Participants Who Underwent Engraftment
Description: Engraftment is the process of transplanted stem cells reproducing new cells.
Time Frame: From randomization until death or as assessed up to 2 years post last participant last treatment visit
Population: Intent-to-treat: Participants who were randomized to receive the treatment and who underwent transplantation.
Measure: Number; unit: Participants
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Number analyzed (Participants) | 30 | 28
Participants | 25 | 25

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Thalidomide + Dexamethasone | DOXIL + Thalidomide + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 48/110 | 53/106
Other Adverse Events (participants affected / at risk) | 110/110 | 104/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide + Dexamethasone (N=110) | DOXIL + Thalidomide + Dexamethasone (N=106)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 3
Bundle Branch Block Right (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tongue Disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 3 | 3
Chest Pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Disease Progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Mass (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Bacterial Infection (Infections and infestations) | 0 | 1
Catheter Related Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis Enterococcal (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 7
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Staphylococcal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1
Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Ejection Fraction Decreased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy Steroid (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Sleep Apnoea Syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 5
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 5 | 3
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cryptogenic Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Arthrectomy (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 5 | 4
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide + Dexamethasone (N=110) | DOXIL + Thalidomide + Dexamethasone (N=106)
Anaemia (Blood and lymphatic system disorders) | 21 | 31
Leukopenia (Blood and lymphatic system disorders) | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Cushingoid (Endocrine disorders) | 5 | 7
Vision Blurred (Eye disorders) | 9 | 16
Abdominal Pain (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 45 | 48
Diarrhoea (Gastrointestinal disorders) | 15 | 16
Dry Mouth (Gastrointestinal disorders) | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 10 | 6
Dysphagia (Gastrointestinal disorders) | 3 | 7
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 26 | 39
Stomatitis (Gastrointestinal disorders) | 4 | 14
Vomiting (Gastrointestinal disorders) | 13 | 15
Asthenia (General disorders) | 19 | 13
Fatigue (General disorders) | 58 | 58
Mucosal Inflammation (General disorders) | 4 | 20
Oedema (General disorders) | 12 | 16
Oedema Peripheral (General disorders) | 53 | 60
Pyrexia (General disorders) | 14 | 16
Candidiasis (Infections and infestations) | 3 | 9
Oral Candidiasis (Infections and infestations) | 2 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 14
International Normalised Ratio Increased (Investigations) | 7 | 8
Weight Decreased (Investigations) | 9 | 9
Weight Increased (Investigations) | 7 | 5
Anorexia (Metabolism and nutrition disorders) | 12 | 16
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 10
Dehydration (Metabolism and nutrition disorders) | 10 | 10
Diabetes Mellitus (Metabolism and nutrition disorders) | 7 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 16
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 12 | 10
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14 | 13
Dizziness (Nervous system disorders) | 27 | 23
Dysgeusia (Nervous system disorders) | 10 | 16
Headache (Nervous system disorders) | 18 | 4
Hypoaesthesia (Nervous system disorders) | 16 | 14
Neuropathy (Nervous system disorders) | 13 | 15
Neuropathy Peripheral (Nervous system disorders) | 22 | 17
Paraesthesia (Nervous system disorders) | 16 | 13
Peripheral Sensory Neuropathy (Nervous system disorders) | 14 | 12
Somnolence (Nervous system disorders) | 13 | 2
Tremor (Nervous system disorders) | 20 | 22
Anxiety (Psychiatric disorders) | 16 | 16
Confusional State (Psychiatric disorders) | 8 | 4
Depression (Psychiatric disorders) | 15 | 15
Insomnia (Psychiatric disorders) | 24 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 24
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 11
Erythema (Skin and subcutaneous tissue disorders) | 7 | 7
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 39
Rash (Skin and subcutaneous tissue disorders) | 20 | 20
Deep Vein Thrombosis (Vascular disorders) | 4 | 10
Hypertension (Vascular disorders) | 2 | 9
Hypotension (Vascular disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days